CLINICAL TRIAL: NCT06087640
Title: A Phase 3/3b, Randomized, Observer-blind, Multicenter Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of an MF59-Adjuvanted Subunit Inactivated Influenza Vaccine Compared to a Non-adjuvanted Influenza Vaccine in Adults ≥65 Years of Age
Brief Title: A Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of an Adjuvanted Influenza Vaccine Compared to a Non-adjuvanted Influenza Vaccine in Adults ≥65 Years of Age
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V118_24
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Influenza, Human
Keywords: Influenza; Vaccine; MF59 adjuvant; aQIV; aTIV; A/H1N1; A/H3N2; B/Yamagata; B/Victoria
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MF59-adjuvanted influenza vaccine (Experimental): MF59-adjuvanted QIV containing 2 influenza type A strains and 2 influenza type B strains or MF59-adjuvanted TIV containing 2 influenza type A strains and 1 influenza type B strain
  Interventions: Biological: aQIV or aTIV
- Non-adjuvanted influenza vaccine (Other): Non-adjuvanted QIV containing 2 influenza type A strains and 2 influenza type B strains or Non-adjuvanted TIV containing 2 influenza type A strains and 1 influenza type B strain
  Interventions: Biological: QIV or TIV

INTERVENTIONS:
Biological: aQIV or aTIV — Participants receive a 0.5-mL intramuscular dose of aQIV or aTIV on Day 1. A 0.5 mL dose of aQIV contains nominally 15 µg of hemagglutinin (HA) of each of the 2 influenza type A strains and each of the 2 influenza B strains (total of 60 µg HA). A 0.5 mL dose of aTIV contains nominally 15 µg of HA of each of the 2 influenza type A strains and of the influenza B strain (total of 45 µg HA). The strain composition of aQIV and aTIV is that recommended by the World Health Organization (WHO) for quadrivalent and trivalent influenza vaccines, respectively, contemporaneous to the timing of the study.
  Other Names: Fluad Tetra/Quadrivalent or Fluad
  Arms: MF59-adjuvanted influenza vaccine
Biological: QIV or TIV — Participants receive a 0.5-mL intramuscular dose of the non-adjuvanted QIV or TIV on Day 1. A 0.5 mL dose of QIV contains nominally 15 μg of HA of each of the 2 influenza type A strains and each of the 2 influenza B strains (total of 60 μg HA). A 0.5 mL dose of TIV contains nominally 15 μg of HA of each of the 2 influenza type A strains and of the influenza B strain (total of 45 μg HA). The strain composition of QIV and TIV is that recommended by the WHO for quadrivalent and trivalent influenza vaccines, respectively, contemporaneous to the timing of the study.
  Arms: Non-adjuvanted influenza vaccine

SUMMARY:
This Phase 3 study is a randomized, observer-blind study of MF59-adjuvanted influenza vaccine (aQIV or aTIV) compared with a non-adjuvanted influenza vaccine (QIV or TIV) in adults ≥65 years of age. The aim of the study is to evaluate MF59-adjuvanted influenza vaccine compared with non-adjuvanted influenza vaccine in the prevention of reverse transcription-polymerase chain reaction (RT-PCR)-confirmed influenza A and/or B in subjects ≥65 years of age.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

1. Adults of ≥65 years of age on the day of vaccination.
2. Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who have the ability to comply with study procedures including follow-up.

Exclusion Criteria:

In order to participate in this study, all subjects must not meet any of the exclusion criteria described below:

1. Bedridden subjects (i.e. confined to bed by sickness or old age).
2. Subjects that are incapacitated and because of that in need of a Legally Authorized Representative.
3. Receipt of any influenza vaccine within 6 months prior to enrollment or any plan to receive influenza vaccine while participating in the study.
4. Hypersensitivity, including allergy, to any component of vaccines whose use is foreseen in this study, or severe allergic reaction (e.g. anaphylaxis) to previous influenza vaccination.
5. Known history of Guillain-Barré syndrome or another demyelinating disease such as encephalomyelitis and transverse myelitis.
6. Clinical conditions representing a contra-indication to intramuscular administration of vaccines or blood draw.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions;
   2. Systemic administration of corticosteroids (PO/IV/IM) at a dose ≥20 mg/day of prednisone (or equivalent) for more than 14 consecutive days within 90 days prior to informed consent; Topical, inhaled and intranasal corticosteroids are permitted. Intermittent use (one dose in 30 days) of intra-articular corticosteroids are also permitted;
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Receipt of immunoglobulins or any blood products within 180 days prior to informed consent.
9. Receipt of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the study vaccination, or planned use during the entire study period.
10. Acute (severe) febrile illness.
11. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
12. Study personnel or immediate family members (brother, sister, child, parent) or the spouse of study personnel.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35800 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint: First-occurrence of RT-PCR-confirmed influenza, due to any influenza Type A and/or B virus (regardless of antigenic match), using the protocol-defined ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for Northern Hemisphere [NH] influenza season and end of November for Southern Hemisphere [SH] influenza season)
  ILI = influenza-like illness; RT-PCR = reverse transcription-polymerase chain reaction

SECONDARY OUTCOMES:
Efficacy Endpoint: First-occurrence of influenza, due to influenza Type A and/or B virus antigenically matched to the vaccine strains selected for the seasonal vaccine, using the protocol-defined ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for NH influenza season and end of November for SH influenza season)
Efficacy Endpoint: First-occurrence of culture-confirmed influenza, due to any influenza Type A and/or B virus (regardless of antigenic match), using the protocol-defined ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for NH influenza season and end of November for SH influenza season)
Efficacy Endpoint: First-occurrence of RT-PCR-confirmed influenza, due to any influenza Type A and/or B virus (regardless of antigenic match), using the modified CDC ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for NH influenza season and end of November for SH influenza season)
  CDC = Centers for Disease Control and Prevention
Efficacy Endpoint: First-occurrence of RT-PCR-confirmed influenza, due to any influenza Type A and/or B virus (regardless of antigenic match), using the WHO ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for NH influenza season and end of November for SH influenza season)
  WHO = World Health Organization
Efficacy Endpoint: First-occurrence of influenza, due to influenza Type A and/or B virus antigenically unmatched to the vaccine strains selected for the seasonal vaccine, using the protocol-defined ILI definition | From 14 days after vaccination (ie study day 15) and until the end of influenza season (typically end of May for NH influenza season and end of November for SH influenza season)
Immunogenicity Endpoint: Pre- and post-vaccination hemagglutination inhibition (HI) geometric mean titers (GMTs) for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains | Day 1 and Day 22
Immunogenicity Endpoint: GMT ratios (adjuvanted/non-adjuvanted) at Day 1 and Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains | Day 1 and Day 22
Immunogenicity Endpoint: Geometric mean fold increase (GMFI, Day 22/Day1) for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains | Day 1 and Day 22
Immunogenicity Endpoint: Percentage of subjects achieving seroconversion for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains | Day 1 and Day 22
  Seroconversion is defined as the percentage of subjects with either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a ≥4-fold increase in post-vaccination titer.
Immunogenicity Endpoint: Percentage of subjects with HI titer ≥1:40 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains | Day 1 and Day 22
Safety Endpoint: All adverse events (AEs) reported within 30 minutes after vaccination | Day 1
Safety Endpoint: Serious adverse events (SAEs) reported during the entire study period | Day 1 to Day 181 or the end of the influenza season, whichever is longer
Safety Endpoint: Adverse events of special interest (AESIs) reported during the entire study period | Day 1 to Day 181 or the end of the influenza season, whichever is longer
Safety Endpoint: AEs leading to premature withdrawal from the study during the entire study period | Day 1 to Day 181 or the end of the influenza season, whichever is longer

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (254):
- United States (111):
  - 84046-Accel Research Sites - Birmingham, Birmingham, Alabama
  - 84075-Cullman Clinical Trials, Cullman, Alabama
  - 84112-DM Clinical Research - Phoenix, Phoenix, Arizona
  - 84114-Scottsdale Clinical Trials, Scottsdale, Arizona
  - 84045-Lynn Institute of the Ozarks, Little Rock, Arkansas
  - 84070-Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - 84101-West Coast Research LLC, Dublin, California
  - 84124-Leading Edge Research, Encino, California
  - 84104-Zillan Clinical Research, Inglewood, California
  - 84105-Eximia Research - CA, La Mesa, California
  - 84107-Long Beach Research Institute, Long Beach, California
  - 84109-Long Beach Clinical Trials, Long Beach, California
  - 84115-Central Valley Research, Modesto, California
  - 84120-Paradigm Research, Redding, California
  - 84119-Apex Clinical Research, San Diego, California
  - 84125-Lynn Institute of Denver, Aurora, Colorado
  - 84110-Tekton Research, Longmont, Colorado
  - 84123-Paradigm Research, Wheat Ridge, Colorado
  - 84085-Clinical Research Consulting, LLC, Milford, Connecticut
  - 84017-Chase Medical Research, LLC, Waterbury, Connecticut
  - 84029-Imagine Research of Palm Beach County, Boynton Beach, Florida
  - 84067-Innovative Research of West Florida, Inc., Clearwater, Florida
  - 84006-Nature Coast Clinical Research - Crystal River, Crystal River, Florida
  - 84012-Evolution Clinical Trials, Doral, Florida
  - 84016-USA and International Research Inc., Doral, Florida
  - 84061-Velocity Clinical Research - New Smyrna Beach, Edgewater, Florida
  - 84065-Fleming Island Center for Clinical Research, Fleming Island, Florida
  - 84027-SIMEDHealth, LLC, Gainesville, Florida
  - 84019-Green Leaf Clinical Trials, Jacksonville, Florida
  - 84026-Health Awareness, Inc., Jupiter, Florida
  - 84071-3SYNC Research, Lake Worth, Florida
  - 84083-Accel Research Sites Network - St. Petersburg-Largo, Largo, Florida
  - 84082-Global Health Research Center, Inc., Miami Lakes, Florida
  - 84081-Suncoast Research Associates, LLC, Pembroke Pines, Florida
  - 84024-St. Johns Center for Clinical Research, Saint Augustine, Florida
  - 84051-Precision Clinical Research, Sunrise, Florida
  - 84008-Global Health Research Center, Inc. - Tampa, Tampa, Florida
  - 84037-Eximia Research - GA, Atlanta, Georgia
  - 84086-Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - 84054-Centricity Research Columbus, Columbus, Georgia
  - 84013-M3 Wake Research/Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - 84069-Velocity Clinical Research - Savannah, Savannah, Georgia
  - 84039-North Georgia Clinical Research, Woodstock, Georgia
  - 84118-Velocity Clinical Research - Boise, Meridian, Idaho
  - 84060-Great Lakes Clinical Trials LLC, dba Flourish Research, Chicago, Illinois
  - 84022-DM Clinical Research - River Forest, Melrose Park, Illinois
  - 84025-Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - 84042-Velocity Clinical Research - Sioux City, Sioux City, Iowa
  - 84055-Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - 84088-Velocity Clinical Research - Covington, Covington, Louisiana
  - 84052-Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - 84064-Benchmark Research, Metairie, Louisiana
  - 84005-DM Clinical Research - Brookline, Brookline, Massachusetts
  - 84002-ActivMed Practices and Research, LLC, Methuen, Massachusetts
  - 84044-Clarkston Medical Group, Clarkston, Michigan
  - 84018-Quest Research Institute, Farmington Hills, Michigan
  - 84032-Bioscope Clinical Research, LLC, Farmington Hills, Michigan
  - 84001-Revival Research Institute, LLC, Southfield, Michigan
  - 84074-DM Clinical Research - Southfield, Southfield, Michigan
  - 84023-Velocity Clinical Research - Gulfport, Gulfport, Mississippi
  - 84038-Kansas City Research Institute, Kansas City, Missouri
  - 84057-Sundance Clinical Research, St Louis, Missouri
  - 84108-Boeson Research MSO, Missoula, Montana
  - 84030-Velocity Clinical Research - Grand Island, Grand Island, Nebraska
  - 84040-Velocity Clinical Research - Norfolk, Norfolk, Nebraska
  - 84007-Velocity Clinical Research - Omaha, Omaha, Nebraska
  - 84117-M3 Wake Research/CRCN, Las Vegas, Nevada
  - 84103-Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - 84111-Vector Clinical Trials, Las Vegas, Nevada
  - 84106-Las Vegas Clinical Trials, North Las Vegas, Nevada
  - 84003-DM Clinical Research - New Jersey, Jersey City, New Jersey
  - 84122-Albuquerque Clinical Trials, Albuquerque, New Mexico
  - 84048-Velocity Clinical Research - Binghamton, Binghamton, New York
  - 84077-Velocity Clinical Research - Syracuse, East Syracuse, New York
  - 84014-Asheville Clinical Research, Asheville, North Carolina
  - 84089-Velocity Clinical Research - Durham, Durham, North Carolina
  - 84035-Monroe Biomedical Research, Monroe, North Carolina
  - 84102-Eximia Research - NC, Raleigh, North Carolina
  - 84020-M3 Wake Research/Raleigh Clinical Research, LLC, Raleigh, North Carolina
  - 84004-TMA Headlands LLC, dba Trial Management Associates, Wilmington, North Carolina
  - 84079-Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - 84021-Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - 84034-CTI Clinical Research Center, Cincinnati, Ohio
  - 84063-Velocity Clinical Research - Cincinnati (Mt. Auburn), Cincinnati, Ohio
  - 84078-Tekton Research, Yukon, Oklahoma
  - 84121-Velocity Clinical Research - Medford, Medford, Oregon
  - 84050-3SYNC Research, Pittsburgh, Pennsylvania
  - 84009-Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - 84010-M3 Wake Research/Charleston Clinical Trials, LLC, Charleston, South Carolina
  - 84043-Velocity Clinical Research - Gaffney, Gaffney, South Carolina
  - 84056-Coastal Carolina Research Center, LLC, North Charleston, South Carolina
  - 84047-Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - 84053-Velocity Clinical Research - Union, Union, South Carolina
  - 84068-WR-ClinSearch, LLC, Chattanooga, Tennessee
  - 84090-Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - 84084-Clinical Research Associates, Inc., Nashville, Tennessee
  - 84072-WR-Global Medical Research, LLC, Dallas, Texas
  - 84028-Benchmark Research, Fort Worth, Texas
  - 84015-Trio Clinical Trials LLC, Houston, Texas
  - 84062-Activian Clinical Research, Kingwood, Texas
  - 84080-ACRC Trials, Plano, Texas
  - 84031-North Texas Family Medicine, Plano, Texas
  - 84066-Research Your Health, Plano, Texas
  - 84011-Clinical Trials of Texas, LLC, dba Flourish Research, San Antonio, Texas
  - 84076-DM Clinical Research - San Antonio, San Antonio, Texas
  - 84059-DM Clinical Research - Sugar Land, Sugar Land, Texas
  - 84087-DM Clinical Research - Tomball, Tomball, Texas
  - 84049-Charlottesville Medical Research, Charlottesville, Virginia
  - 84058-Clinical Research Partners, Richmond, Virginia
  - 84036-Velocity Clinical Research - Suffolk, Suffolk, Virginia
  - 84113-DM Clinical Research - Seattle, Seattle, Washington
- Australia (14):
  - 03603-University of the Sunshine Coast, Birtinya
  - 03609-Paratus Clinical Western Sydney, Blacktown
  - 03605-Emeritus Research - Sydney, Botany
  - 03614-Northern Beaches Clinical Research, Brookvale
  - 03602-Emeritus Research - Melbourne, Camberwell
  - 03615-Momentum Clinical Research Darlinghurst, Darlinghurst
  - 03608-Paratus Clinical Brisbane, Herston
  - 03610-Paratus Clinical Central Coast, Kanwal
  - 03604-Doherty Clinical Trials Limited, Melbourne
  - 03611-Nucleus Network, Melbourne
  - 03601-University of the Sunshine Coast - Morayfield, Morayfield
  - 03607-University of the Sunshine Coast - South Bank, South Brisbane
  - 03613-Momentum Clinical Research Taringa, Taringa
  - 03612-Wollongong Clinical Reserach, Wollongong
- Belgium (4):
  - 05605-AZ Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges
  - 05602-Universitair Ziekenhuis Gent, Ghent
  - 05603-Medif BVBA, Gozée
  - 05601-Jan Yperman Ziekenhuis, Ieper
- Bulgaria (21):
  - 10005-MHAT Dr. Tota Venkova, Gabrovo
  - 10018-Medical Center - Zdrave-1, Kozloduy
  - 10029-Medical Centre Leo Clinic EOOD, Lovech
  - 10007-Medical Center Hera EOOD, Montana
  - 10014-Multi-Profile Hospital For Active Treatment Dr. Stamen Iliev AD, Montana
  - 10032-MHAT Zdrave, Pazardzhik
  - 10019-MC Med Consult Pleven, Pleven
  - 10022-Ambulatory Outpatient Medical Practice for First Patient Care Zaprin Pepelov, Plovdiv
  - 10024-UMHAT Pulmed, Plovdiv
  - 10026-Multiprofile Hospital for Active Treatment Sv. Panteleymon - Plovdiv, Plovdiv
  - 10031-Medical Centre Pratia Clinic EOOD, Plovdiv
  - 10004-Medical Center Prolet EOOD, Rousse
  - 10012-Specialized Hospital For Active Treatment Of Pneumo-Phthisiatric Diseases Dr. Dimitar Gramatikov-Ruse EOOD, Rousse
  - 10016-Medical Center 1 - Sevlievo EOOD, Sevlievo
  - 10023-DCC-1 Sliven, Sliven
  - 10006-DCC 22 - Sofia, Sofia
  - 10015-Medical Center Hera - Pulmonology Office, Sofia
  - 10021-Medical Center Intermedica, Sofia
  - 10028-Medical Center Excelsior OOD, Sofia
  - 10030-Diagnostic-Consultative Centre Ascendent EOOD, Sofia
  - 10027-AIPPMP D-r Zhaneta Demireva, Stamboliyski
- Czechia (8):
  - 20307-CCR Brno s.r.o., Brno
  - 20305-Centrum ockovani a cestovni mediciny, České Budějovice
  - 20306-ADMED, s.r.o., České Budějovice
  - 20311-Ordinace Hradebni s.r.o, České Budějovice
  - 20310-MUDr. Jakub Strincl, s.r.o., Liberec
  - 20309-CCR Ostrava, s.r.o., Ostrava
  - 20308-MUDr. Jakub Strincl, s.r.o., Protivín
  - 20312-MEDISON s.r.o., Přeštice
- Finland (4):
  - 24603-Helsinki South Vaccine Research Clinic, Helsinki
  - 24602-Oulu Vaccine Research Clinic, Oulu
  - 24601-Tampere Vaccine Research Clinic, Tampere
  - 24604-Turku Vaccine Research Clinic, Turku
- Georgia (4):
  - 26803-UNIMED Adjara LTD - Batumi Referral Hospital, Batumi
  - 26801-LTD Hospital Service, Kutaisi
  - 26802-Acad. G. Chapidze Emergency Cardiology Center, Tbilisi
  - 26804-K. Eristavi National Center of Clinical Surgery, Tbilisi
- Italy (3):
  - 38003-Policlinico Bari, Bari
  - 38001-PO A. Manzoni di Lecco, ASST Lecco, Lecco
  - 38004-Ospedale Fatebenefratelli e Oftalmico, ASST Fatebenefratelli Sacco, Milan
- Lithuania (4):
  - 44004-JSC InMedica, Kaunas
  - 44008-JSC Saulės Šeimos Medicinos Centras, Kaunas
  - 44009-Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - 44010-InlitaJSC Santara CTC, Vilnius
- Netherlands (2):
  - 52802-Emotional Brain BV, Almere Stad
  - 52804-Universitair Medisch Centrum (UMC) Utrecht - Julius Center for Health Sciences and Primary Care, Utrecht
- New Zealand (5):
  - 55404-Optimal Clinical Trials - Central, Grafton
  - 55402-Momentum Clinical Research Wellington, Mount Cook
  - 55405-Pacific Clinical Research Network - West Auckland, New Lynn
  - 55403-Optimal Clinical Trials - North, Rosedale
  - 55401-PCRN - Auckland, Takapuna
- Philippines (14):
  - 60812-Health Index Multispecialty and Lying-In Clinic, Bacoor
  - 60813-Norzel Medical and Diagnostic Clinic, Cebu
  - 60808-CT CARE Group, Dasmariñas
  - 60801-Davao Doctors Hospital, Davao City
  - 60802-West Visayas State University Medical Center, Iloilo City
  - 60815-St Paul's Hospital Iloilo, Iloilo City
  - 60816-St Paul's Hospital Iloilo, Iloilo City
  - 60803-Philippine General Hospital, Manila
  - 60811-Philippine General Hospital, Manila
  - 60814-Manila Doctors Hospital, Manila
  - 60804-St. Michael Family Hospital, Marilao
  - 60805-San Juan de Dios Hospital, Pasay
  - 60806-Quirino Memorial Medical Center, Quezon City
  - 60817-Silang Specialist Medical Center, Silang
- Poland (11):
  - 61619-Krakowskie Centrum Medyczne Sp. z o.o, Krakow
  - 61618-Centrum Medyczne AMED Oddzial w Lodzi, Lodz
  - 61622-KOMED Nova Lublin II, Lublin
  - 61620-KOMED Nova Pulawy, Puławy
  - 61614-KO-MED Centra Kliniczne Staszow, Staszów
  - 61605-RCMed Oddział Warszawa, Warsaw
  - 61615-ETG Warszawa, Warsaw
  - 61616-MTZ Clinical Research, Warsaw
  - 61621-Futuremed Warszawa Centrum, Warsaw
  - 61617-Przychodnia FutureMeds Wroclaw, Wroclaw
  - 61623-KOMED Nova Zamosc, Zamość
- Romania (5):
  - 64210-Sana Monitoring, Bucharest
  - 64208-Spitalul Municipal Caracal, Caracal
  - 64204-Ames Research Center, Călăraşi
  - 64209-Clintrial Medical Center, Reșca
  - 64211-Nova-Clin Medical Research Center, Timișoara
- Serbia (5):
  - 68803-Clinical Center of Serbia, Belgrade
  - 68805-Clinical Hospital Center Zemun, Belgrade
  - 68806-CHC Bezanijska Kosa, Belgrade
  - 68802-Institute for Pulmonary Disease of Vojvodina, Kamenitz
  - 68804-General Hospital Valjevo, Valjevo
- South Africa (12):
  - 71007-Josha Research Center, Bloemfontein
  - 71008-Madibeng Centre for Research, Brits
  - 71011-University of Cape Town Lung Institute, Cape Town
  - 71014-TREAD Research, Cape Town
  - 71015-Tiervlei Trial Centre, Cape Town
  - 71001-Ubuntu Clinical Research Krugersdorp, Krugersdorp
  - 71010-Merclinico Middelburg, Middelburg
  - 71009-Newtown Clinical Research Centre, Newtown
  - 71005-Be Part Research, Paarl
  - 71013-Into Research, Life Groenkloof Hospital, Pretoria
  - 71003-Tsitsikamma Clinical Research Initiative, Thabazimbi
  - 71004-FCRN Clinical Trials Centre, Vereeniging
- South Korea (5):
  - 41002-Korea University Ansan Hospital, Ansan
  - 41001-Inha University Hospital, Incheon
  - 41004-Hallym University Kangnam Sacred Heart Hospital, Seoul
  - 41005-Korea University Guro Hospital, Seoul
  - 41003-Ajou University Hospital, Suwon
- Spain (7):
  - 72402-EAP Vic - CAP El Remei, Barcelona
  - 72407-Futurmeds Spain Cadiz, Cadiz
  - 72405-Futuremeds Spain Madrid, Madrid
  - 72404-Hospital Universitario Son Espases, Palma de Mallorca
  - 72403-Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - 72406-Futuremeds Spain Sevilla, Seville
  - 72401-Hospital Povisa, Vigo
- Taiwan (5):
  - 15803-Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - 15801-China Medical University Hospital, Taichung
  - 15802-National Cheng Kung University Hospital, Tainan
  - 15804-Taipei Medical University - Wanfang Hospital, Taipei
  - 15805-Taipei Medical University, Taipei
- Turkey (Türkiye) (9):
  - 79209-Hacettepe University Faculty of Medicine, Ankara
  - 79207-Akdeniz University Faculty of Medicine, Antalya
  - 79212-Dicle Universitesi Tip Fakultesi, Diyarbakır
  - 79205-Goztepe Suleyman Yalcin City Hospital, Istanbul
  - 791210-Dokuz Eylul University Faculty of Medicine, Izmir
  - 79208-Izmir Dr. Suat Seren Pulmonary Hospital, Izmir
  - 79213-Ege University Hospital, Izmir
  - 79204 - Kocaeli University Faculty of Medicine, Kocaeli
  - 79211-Karadeniz Technical University Faculty of Medicine, Trabzon
- 71601-Charles River Medical Group, Mutala Trust and Infectious Disease Research Laboratory, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Seqirus will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact Seqirus at seqirus.clinicaltrials@seqirus.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.